CLINICAL TRIAL: NCT03344601
Title: A Longitudinal Cohort Study With Nested Randomised Pragmatic Controlled Trial to Evaluate Physical Activity and Exercise Related Outcomes in People With Huntington's Disease
Brief Title: PHysical Activity and Exercise Outcomes in Huntington's Disease
Acronym: PACE-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiff University (Other)
Collaborators: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SPON 1631-17
Record Dates: First submitted 2017-10-17; First posted 2017-11-17 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a 12 month observational study with a nested randomised controlled trial of a physical activity intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference Cohort (No Intervention): A 12-month longitudinal evaluation of physical fitness and physical activity assessments in a cohort of individuals with HD (n=60) recruited from the Enroll-HD platform study.
- Physcial Activity Intervention (Experimental): Participants will be recruited from the Enroll-HD platform study and will be individually randomised (1:1) to a 12-month physical activity and coaching intervention.
  Interventions: Behavioral: physical activity
- Activity as usual control (No Intervention): Participants will be recruited from the Enroll-HD platform study and will be individually randomised (1:1) to continue with physical activity as usual for 12 months

INTERVENTIONS:
Behavioral: physical activity — The program will consist of 18 face-to-face coaching sessions (~1 hour) over 12 months. The timing of these sessions will be decided between participant and coach. A coaching manual will be used to provide a structured approach to coaching sessions, focussing on physical activity engagement (specifically aerobic and strengthening exercise) and adherence to exercise. The intervention will take place in the participant's home or in a rehabilitation facility at the research site. Each participant will be provided with a choice of exercise equipment options (e.g. exercise bike, weights, therabands), gym membership or use of online exercise resources. Participants will develop physical activity goals that will be monitored and adjusted throughout the program. Physical activity diaries will be completed to record the amount and type of physical activity involvement. Wearable activity monitors will also be used to facilitate/monitor physical activity and sedentary behaviours.
  Arms: Physcial Activity Intervention

SUMMARY:
Huntington's disease (HD) is a genetic, degenerative neurological disease that affects individuals in their third-fourth decade of life and individuals can live 15-20 years with manifest HD. The complex disease symptoms, including motor, cognitive and behavioural impairments, result in loss of functional independence and progressive escalation of healthcare costs. The personal, social and economic consequences of HD are devastating, especially as there are currently no disease modification therapies available.

Environmental factors, including exercise and physical activity, have the potential to minimize the functional impact of HD. Animal models of HD have provided the first evidence that exercise has the potential to delay or alter disease progression. A range of studies in clinical populations have shown that short-term exercise (< 3 months) is well tolerated and has the potential to improve quality of life, fitness and motor impairments in HD. Despite these promising studies, there are critical knowledge gaps that prevent the intelligent application of exercise as a therapeutic intervention in HD. Firstly, there have been no prospective evaluations of the potential role of physical activity and exercise in disease modification in HD. To date, only retrospective data has suggested that lifestyle factors, including sedentary behavior, could negatively affect disease progression in HD. Secondly, it is not known if sustained exercise (> 3 months) is feasible, and if it has the potential to improve cognitive outcomes, such as has been shown in other neurodegenerative diseases. Such longer-term studies are essential to elucidate the potential for exercise to have a disease-modifying effect; the mechanisms through which such improvement may occur have yet to be explored.

In this trial, the investigators will employ a systematic approach for routinely collecting prospective physical activity and fitness data and monitoring physical activity behaviour in 120 individuals with HD. The investigators will use a database to track physical activity and exercise behaviour alongside standardized disease-specific outcome measures during two annual visits. Assessment will incorporate VO2max, a surrogate measure of fitness and a direct measure of oxygen uptake related to central nervous system (CNS) function and structure, and the use of wearable technologies (Gene-activ activity monitors) that capture and quantify dose (frequency, duration, intensity) of physical activity in a large HD cohort. The investigators will further conduct a within-cohort randomized control trial (RCT) of a 12-month exercise intervention in HD, comparing a supported structured aerobic exercise training program to activity as usual. This intervention will also incorporate a physical activity coaching program developed and evaluated by our group with a view to encouraging longer term exercise uptake.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a neurodegenerative disease causing dysfunction and death of medium spiny striatal projection neurons and thus disruption of corticostriatal pathways with resultant impairment of cognition, motor function, and behaviour. These impairments result in decreasing independence in activities of daily living and quality of life even from relatively early in the disease. The potential to develop interventions to facilitate independent living and strategies to manage symptoms is crucial to managing both the personal and economic effects of this devastating disease. Although to date there are no successful pharmacological interventions that are able to slow disease progression, there is now clear emerging evidence of disease specific motor function and general health benefits of shorter exercise in HD. Although it has been possible to successfully deliver exercise and behaviour change interventions in HD over the shorter term, there is now a need to conduct studies that actively facilitate exercise adherence over a longer term (e.g. one year) to realistically begin to assess the impact of physical activity and structured exercise on disease progression.

Therapeutic exercise interventions present an exciting, transformative area of research in neurodegenerative diseases. Addressing motor impairments in neurodegeneration may provide a long-term beneficial effect in delaying disease progression and maximizing functional abilities over a longer period. Loss of independent mobility and care dependency have been shown to be important predictors of nursing home admissions. The potential to develop interventions that facilitate independent living and strategies to manage symptoms is crucial to managing both the personal and economic effects of this devastating disease. Although to date there are no successful pharmacological or other interventions that are able to slow disease progression, there is some suggestion that lifestyle factors, such as activity level and education alongside specific motor training may help to drive compensatory neural networks, that may in turn compensate for the failing brain, and change the course of the disease. Studies to date in HD have relied on retrospective data, and robust evaluation of lifestyle factors contributing to disease progression is needed. If shown to be effective, exercise programs have the potential to be used in combination with disease-modifying drugs, cell replacement therapy or genetic manipulations, when available, to maximize the functional benefits of these interventions by facilitating adaptive neuroplasticity.

The investigators have set out to systematically evaluate the feasibility of exercise and physical activity interventions in people with HD using a two-pronged approach. The first approach evaluated the feasibility of short-term aerobic and strengthening exercise programs in HD. This led to the recently completed study funded by the Gossweiler Foundation, Exert-HD, a 3-month randomized controlled trial of aerobic (performed between 60-85% age predicted heart rate max) and strengthening exercise. Participants in the exercise group demonstrated significantly improved predicted VO2 max and Unified Huntington Disease Rating Scale (UHDRS) modified Motor Scores (mMS), but no effect was seen on cognition or other measures of motor function.This study had high retention and adherence, and was well tolerated by participants. Alongside this, there was the development and evaluation of the feasibility of a behavioural change intervention to increase levels of physical activity (Engage-HD; ISRCTN65378754). The intervention aimed to evaluate the efficacy of a physical activity intervention (6 sessions over 14 weeks) utilizing a workbook-based behavioural change program compared to a social contact control. This study demonstrated improvements in self-reported physical activity, self-efficacy for exercise, and cognition, however no changes were noted for HD-specific motor function.

In PACE-HD the investigators seek to address three issues that naturally arise from the preliminary studies completed to date. First, there has been no evaluation of long-term (e.g. 12 month) aerobic and strengthening exercise interventions in HD. While studies to date have demonstrated improvements in motor and cognitive function in the short term, it is unclear whether exercise behaviour can be maintained over a longer term, and to what degree any improvements in cognition or motor function can be maintained or enhanced with a longer term intervention.

Second, there is a lack of understanding of the role of physical activity in disease progression in HD. Preliminary work has utilized 7 day activity monitors that have improved functionality to obtain more detailed data on physical activity behavior, including light and moderate- vigorous physical activity, sedentary behavior and sleep patterns over the intervention period. In this trial, the investigators will utilize 7 day activity monitors to evaluate activity patterns longitudinally over a year period in a cohort of 120 people with HD. This longitudinal evaluation alongside standardized evaluations of motor, cognitive and functional abilities will aid in validation of wearable activity devices and evaluate how physical fitness and physical activity may be related to disease progression.

Third, there is lack of understanding of the mechanisms by which exercise may achieve its effect in HD. Trials of longer term exercise interventions are difficult to deliver, not least in terms of the complexity of the intervention but also due to the challenges in accurately characterising the different dimensions of real-life physical activity and understanding individual response to exercise. Our preliminary research has shown that exercise has the potential to improve aerobic fitness using measurements of estimated (predicted) VO2max. This trial will incorporate longitudinal assessment of VO2max, a surrogate measure of fitness and a direct measure of oxygen uptake that is related to central nervous system (CNS) function and structure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD, confirmed by genetic testing
* Above the age of 18
* A participant (current or newly enrolled) in the Enroll-HD study
* Up to and including stage 2 disease status (TFC 7-13)

Exclusion Criteria:

* Diagnosis of juvenile onset HD
* History of co-morbid neurological conditions such as multiple sclerosis or stroke
* Acute orthopaedic conditions (within a month) e.g. ankle sprain or fracture
* Inability or unwillingness of participant or legal guardian to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Data completeness | 12 months
  The amount of trial data completed will be recorded. The amount of complete data will be analysed in reference to the amount of data expected for each participant to give a percentage score of data completeness for each participant. This will give an over percentage data completion rate for the whole trial. The percentage of complete data will be looked at in combination with measures of recruitment, retention, safety, adherence, fidelity and acceptability to assess the overall feasibilty of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Recruitment | 12 months
  Recruitment to target within the pre-defined recruitment period of 9 months will be recorded. This will result in a percentage value of recruitment to target and will be looked at in combination with measures of data completeness, retention, safety, adherence, fidelity and acceptability to assess the overall feasibilty of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Retention | 12 months
  The retention of participants to the trial will be recorded. The number of participants who actually complete the trial will be compared to the number of participants in the intervention arm expected to complete the trial will be used to determine the percentage retention of participants and will be used in combination with measures of data completeness, recruitment, safety, adherence, fidelity and acceptability to assess the overall feasibilty of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Safety | 12 months
  All adverse events in the intervention and comparator arms of the nested RCT will be recorded.The total number of adverse events in each arm will be analysed to see if there is a signifcant difference in the number of events between the two arms. Any difference in the number of adverse events between arms will be used in combination with measures of data completeness, recruitment, retention, adherence, fidelity and acceptability to assess theoverall feasibilty of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Adherence | 12 months
  The adherence of participants to the intervention will be measured using self report diaries and automated activity monitors. These will be analysed to ensure the participants have adhered to the intervention to an acceptable level. The level of adherence of individual participants will be combined to generate an overall percentage adherence score and this will be used in combination with measures of data completeness, recruitment, retention, safety, fidelity and acceptability to assess the feasibility of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Fidelity | 12 months
  The fidelity of the intervention delivery by therapists will be assessed through the monitoring of three coaching sessions with each participant. Each monitored session will be analysed and scored on a scale of 0-4 (with 0 = not at all and 4=to a great extent) across 4 domains to give an overall score (maximum 16). Fidelity scores for each participant/ coach will be used to generate on overall fidelity score and this will be used in combination with measures of data completeness, recruitment, retention, safety, adherence and acceptability to assess the feasibility of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.
Acceptability | 12 months
  The acceptability of the intervention to participants will be assessed in a post-study questionnaire about specific aspects of the intervention and taking part in the trial. The questionnaire will be a combination of answers using a likert scale from 1-5 (1= strongly agree, 5=strongly agree) and free text responses. Quantitative analysis of the responses will give an overall acceptability score per participant which will be used to produce an average accepatability score. This and qualitative analysis of the free text responses will be used in combination with measures of data completeness, recruitment, retention, safety, adherence and fidelity to assess the feasibility of the trial. The trial will be determined to be feasible if the majority of components investigated reach pre-determined criteria.

SECONDARY OUTCOMES:
Work rate (measured in Watts) | Baseline, 6 months (RCT only), 12 months
  This will be measured during stepwise incremental exercise test. The test is performed on a cycle ergometer with participants seated in a standardized position. Participants will attempt to maintain a cadence of 50 revolutions per minute (rpm), starting at 50 Watts and increasing by 25 Watts every two minutes until test termination. The test will be terminated when the participant reaches volitional exhaustion or cadence drops by 10 rpm. At the end of each increment, work-rate (Watts), This will be used with the rating of perceived exertion and heart rate to calculate the predicted VO2 max.
Rating of perceived exertion (Borg RPE scale) | Baseline, 6 months (RCT only), 12 months
  This will be measured during stepwise incremental exercise test. The test is performed on a cycle ergometer with participants seated in a standardized position. Participants will attempt to maintain a cadence of 50 revolutions per minute (rpm), starting at 50 Watts and increasing by 25 Watts every two minutes until test termination. The test will be terminated when the participant reaches volitional exhaustion or cadence drops by 10 rpm. At the end of each increment rating of perceived exertion using the Borg RPE scale (where participants rate their effort on a scale of 1 [very light activity] to 10 [maximal effort activity]). This will be used with Watts and heart rate to calculate the predicted VO2 max.
Heart Rate (beats per minute) | Baseline, 6 months (RCT only), 12 months
  This will be measured during stepwise incremental exercise test. The test is performed on a cycle ergometer with participants seated in a standardized position. Participants will attempt to maintain a cadence of 50 revolutions per minute (rpm), starting at 50 Watts and increasing by 25 Watts every two minutes until test termination. The test will be terminated when the participant reaches volitional exhaustion or cadence drops by 10 rpm. At the end of each increment heart rate will be recorded for analysis will be used with Watts and rating of perceived exertion to calculate the predicted VO2 max.
Predicted VO2 Max | Baseline, 6 months (RCT only), 12 months
  This will be measured during stepwise incremental exercise test. The test is performed on a cycle ergometer with participants seated in a standardized position. Participants will attempt to maintain a cadence of 50 revolutions per minute (rpm), starting at 50 Watts and increasing by 25 Watts every two minutes until test termination. The test will be terminated when the participant reaches volitional exhaustion or cadence drops by 10 rpm. At the end of each increment, work-rate (Watts), rating of perceived exertion (Borg RPE scale) and heart rate will be recorded for analysis and conversion to predicted VO2 max score.
6 minute walk | Baseline, 6 months (RCT only) and 12 months
  The 6-minute walk test will be used as a measure of walking endurance. This test evaluates the distance walked over a 6 minute period, and has been validated for use in HD.
HD Pro-Triad | Baseline and 12 months
  This will be used to assess disease specific symptoms including cognitive decline, emotional/behavioural dyscontrol and motor dysfunction.
Brunel Lifestyle Physical Activity Questionnaire | Baseline, 6 months (RCT only) and 12 months
  This is a self-report instrument that measures the planned and unplanned dimensions of lifestyle physical activity.
Gene-activ assessment | Baseline, 6 months (RCT only) and 12 months
  Research-grade physical activity monitors (Gene-activs) will be used for a 7-day physical activity assessment. Participants will be given the monitors at the consent visit, and will be asked to return them at the baseline visit one week later. They will be requested to wear them for 24 hours a day for the full week, except when showering. Participants will be given the monitors at the end of the assessments, and will be given addressed stamped mailing envelopes to return the monitors one-week later. Data obtained for analysis will include level of overall physical activity, sedentary behavior and sleep patterns.
International Physical Activity Questionnaire (Short Form) | Baseline, 6 months (RCT only) and 12 months
  This will be used to assess 7-day physical activity, and to validate with the physical activity monitors
The Clinch Token Transfer Test (C3T) | Baseline and 6 months
  [RCT sites only] This is a dual-task assessment of bilateral, upper motor function that consists of three-coin transfer tasks which increase in difficulty (baseline simple, baseline complex and a dual task). The time taken to pick up and transfer the coins from dominant to non-dominant hand and place into a purpose developed box is recorded. The addition of cognitive load increases the task complexity.
Q Motor | Baseline and 12 months
  [RCT sites only] This was developed in TRACK-HD and TRACK-ON-HD where motor tasks are related to functionally relevant everyday tasks. All Q-Motor assessments are based on the application of pre-calibrated and temperature controlled force transducers and 3D position sensors with very high sensitivity and test-retest reliability across sessions and sites in a multicenter clinical trial.
Lorig Self Efficacy | Baseline, 6 months (RCT only) and 12 months
  [RCT sites only] The Lorig scale measures self efficacy in people with chronic disease. Specifically the exercise sub-domain will be measured. Participants are asked to rate their confidence from 1 (not at all confident) to 10 (totally confident) against 3 questions related to undertaking exercise. The scores for each question are summated to give an average score.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Busse, PhD, Principal Investigator — Cardiff University; Lori Quin, PhD, Principal Investigator — Teacher's College, Columbia University
Locations (6):
- United States (2):
  - Re+Active Therapy and Wellness Centre/ UCLA, Los Angeles, California
  - Teacher's College, Columbia University, New York, New York
- Germany (2):
  - George Huntington Institute, Münster
  - University Hospital Ulm, Ulm
- Spain (2):
  - Merce de Deu de la Mare, Barcelona
  - Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The final study data will be shared with the CHDI Foundation Inc.
Time Frame: Data will become available at the conclusion of the study after the primary study results have been published in an open acces journal.
Access Criteria: Applications for the dta must be made to CHDI

REFERENCES:
- [Derived] Quinn L, Playle R, Drew CJG, Taiyari K, Williams-Thomas R, Muratori LM, Hamana K, Griffin BA, Kelson M, Schubert R, Friel C, Morgan-Jones P, Rosser A, Busse M; PACE-HD site investigators. Physical activity and exercise outcomes in Huntington's disease (PACE-HD): results of a 12-month trial-within-cohort feasibility study of a physical activity intervention in people with Huntington's disease. Parkinsonism Relat Disord. 2022 Aug;101:75-89. doi: 10.1016/j.parkreldis.2022.06.013. Epub 2022 Jun 29. PMID 35809488
- [Derived] Drew CJG, Quinn L, Hamana K, Williams-Thomas R, Marsh L, Dimitropoulou P, Playle R, Griffin BA, Kelson M, Schubert R, Muratori L, Reilmann R, Rosser A, Busse M. Physical Activity and Exercise Outcomes in Huntington Disease (PACE-HD): Protocol for a 12-Month Trial Within Cohort Evaluation of a Physical Activity Intervention in People With Huntington Disease. Phys Ther. 2019 Sep 1;99(9):1201-1210. doi: 10.1093/ptj/pzz075. PMID 31101920
- [Derived] Rodrigues FB, Quinn L, Wild EJ. Huntington's Disease Clinical Trials Corner: January 2019. J Huntingtons Dis. 2019;8(1):115-125. doi: 10.3233/JHD-190001. PMID 30776019